CLINICAL TRIAL: NCT06030011
Title: Implementing the NYU Electronic Patient Visit Assessment (ePVA) for Head and Neck Cancer In Rural and Urban Populations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Cancer Institute (NCI) (NIH); New York University Meyers College of Nursing (Unknown); New York University Langone Perlmutter Cancer Center (Unknown); University of Kansas (Other); Fox Chase Cancer Center (Other)
Responsible Party: Principal Investigator, Janet Van Cleave, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-SN-23-0784
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NYU Electronic Patient Visit Assessment (ePVA) plus Usual Care (Experimental)
  Interventions: Behavioral: NYU Electronic Patient Visit Assessment (ePVA); Behavioral: Usual Care
- Usual Care (Active Comparator)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: NYU Electronic Patient Visit Assessment (ePVA) — The NYU Electronic Patient Visit Assessment (ePVA) for head and neck cancer is a digital patient-reported symptom monitoring system, providing actionable information at point-of-care that enables clinicians to provide real-time interventions. Patients access the ePVA through a web link and complete the survey questions within 10 minutes on digital devices (e.g., smart phones, laptops, or digital devices provided by the clinic).
  Arms: NYU Electronic Patient Visit Assessment (ePVA) plus Usual Care
Behavioral: Usual Care — Usual care encompasses pre-treatment, on treatment, and post-treatment care. Pre-treatment care includes education of patients on the treatment plan. On-treatment care includes daily monitoring by a nurse in the radiation therapy (RT) department, weekly on-treatment visits with the RT nurse practitioner and radiation oncologist, and weekly visits with medical oncology nurse practitioners and medical oncologists for patients receiving RT plus chemotherapy. Post-treatment care includes follow-up visits with HNC clinicians (i.e., surgeon, medical oncologist, oral maxillofacial surgeons, and radiation oncologist) to assess the patient's cancer status and identify the patient's acute and long-term symptoms. The clinician's decisions on radiologic exams and referrals to appropriate specialist services, including dental care, are based on the patient's cancer status and symptoms.

SUMMARY:
The PI and the research team developed the New York University (NYU) Electronic Patient Visit Assessment (ePVA) for head and neck cancer (HNC) as a patient-reported outcome measure (PRO) for the early detection of uncontrolled symptoms. The ePVA is digital patient-reported symptom monitoring system, providing actionable information at point-of-care that enables clinicians to provide real-time interventions. The study aims to advance the science of cancer care delivery by testing the effectiveness of the ePVA as a digital patient-reported monitoring system for patients with HNC in real-world settings and identify implementation strategies that optimize the effectiveness of the ePVA in diverse rural and urban settings. The study hypothesis is that participants assigned to the ePVA arm will have better swallowing, taste and smell, and social function than participants assigned to usual care arm at 4 weeks after completing radiation therapy.

ELIGIBILITY:
Inclusion Criteria (Patient Participants):

* Individuals with histologically diagnosed head and neck cancer (HNC) undergoing curative radiation therapy with or without chemotherapy
* English or Spanish speaking

Inclusion Criteria (Clinician Participants):

* Clinicians (i.e., physicians, nurses, dentists, physician assistants, social workers, nutritionists, speech swallow therapists) caring for patients with head and neck cancer at the participating institutions

Exclusion Criteria (Patient and Clinician Participants):

* Any medical condition that could limit the participant's ability to provide informed consent and complete the questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Head and neck cancer (HNC) symptoms as assessed by the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaires (QLQ) | 4 weeks after completing radiation therapy
  The EORTC QLQ-C30 and QLQ-H&N35 will be used to measure head and neck cancer symptoms, such as social function, senses of taste and smell, and swallowing. The scores will be summed and then transformed to a single score ranging from 0=Best to 100=Worst.

SECONDARY OUTCOMES:
Pain as assessed by EORTC QLQ-H&N35 Quality of Life Questionnaire (QLQ) | 4 weeks after completing radiation therapy
  The EORTC QLQ-H&N35 will be used to assess pain. The score will be summed and then transformed to a single score ranging from 0=Best to 100=Worst.
Health-Related Quality of Life (HRQoL) as assessed by the EORTC QLQ-C30 Quality of Life Questionnaire (QLQ) | 4 weeks after completing radiation therapy
  The EORTC QLQ-H&N35 will be used to assess Health-Related Quality of Life (HRQoL). The score will be summed and then transformed to a single score ranging from 0=Best to 100=Worst.
Acute Care Services Use as assessed by number of acute care visits | 4 weeks after completing radiation therapy
  Acute Care Services Use is the use of services delivered in acute care settings, such as feeding tube placements, emergency room visits, and hospitalizations.
Acute Care Services Use as assessed by number of days of using acute care | 4 weeks after completing radiation therapy
  Acute Care Services Use is the use of services delivered in acute care settings, such as feeding tube placements, emergency room visits, and hospitalizations.

CONTACTS AND LOCATIONS:
Overall Officials: Janet H. Van Cleave, PhD, RN, Principal Investigator — The University of Texas Health Science Center at Houston (UTHealth Houston)
Locations (5):
- United States (5):
  - University of Kansas Cancer Center, Kansas City, Kansas
  - NYU Meyers College of Nursing, New York, New York
  - NYU Langone Perlmutter Cancer Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UTHealth Houston Cizik School of Nursing, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van Cleave JH, Brody AA, Schulman-Green D, Hu KS, Li Z, Johnson SB, Major VJ, Lominska CE, Bauman JR, Hanania AN, Tatlonghari GV, Tsikis M, Egleston BL. Implementing the NYU Electronic Patient Visit Assessment (ePVA)(c) for head and neck cancer in rural and urban populations: a study protocol for a type 1 hybrid effectiveness-implementation clinical trial. Trials. 2025 Dec 9;26(1):563. doi: 10.1186/s13063-025-09268-w. PMID 41366462